CLINICAL TRIAL: NCT03404258
Title: ET1 Concentration, Metabolic Pathway Activation, and Pulmonary Blood Flow in Infants Undergoing Superior Cavo-Pulmonary Anastomosis
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0832
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Single-ventricle; Pulmonary Vascular Resistance Abnormality; Superior Cavo-Pulmonary Anastomosis; Endothelin; Metabolomics
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study Patients: Infants between 1 month and 2 years of age undergoing evaluation for SCPA candidacy.
  Interventions: Other: Research Blood Sampling
- Control Patients: Infants between 3 months and 12 months of age with no known cardio-pulmonary disease, no active infection, and no known genetic abnormality undergoing elective surgery for a non-cardiac indication.
  Interventions: Other: Research Blood Sampling

INTERVENTIONS:
Other: Research Blood Sampling — Blood samples will be collected at specified time points and research assays will be performed.

SUMMARY:
This is a novel preliminary study of biomarkers of pathologic pre-operative pulmonary vascular development, elevated pre-operative Pulmonary Vascular Resistance Index (PVRi), and complications associated with decreased post-operative pulmonary blood flow in single ventricle patients undergoing superior cavo-pulmonary anastomosis (SCPA). The study will utilize a combined targeted and untargeted approach to both optimize translation of a promising existing biomarker and efficiently identify novel biomarkers and potential therapeutic targets in this population.

DETAILED DESCRIPTION:
Overall Hypothesis: Endothelin-1 (ET1) and associated dysregulation of key metabolic pathways decrease pre-operative pulmonary blood vessel development and increase post-operative pulmonary blood vessel resistance leading to decreased pulmonary blood flow in patients undergoing SCPA.

For enrolled patients, collected data will include:

* 3 mL blood sample (x2) at pre-SCPA catheterization.
* 3 mL blood samples at 2, 24, and 48 hours post-operative.
* Urine sample pre-operatively and post-operatively
* Collection of otherwise-discarded operative tissue sample from the pulmonary artery.
* Collection of clinical data, demographic data, and results of routine, post-operative hemodynamic monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease patients undergoing catheterization for pre-SPCA evaluation or undergoing SCPA without plans for cardiac catheterization (utilizing data from a previously performed clinical catheterization).
* All patients will have age from 31 days to 2 years.

Exclusion Criteria:

* Patients who will remain post-op with a pulsatile source of pulmonary blood flow in addition to the cavo-pulmonary anastomosis (so called "1.5 ventricle" repair) will be excluded.
* Due to limitations in acceptable sample blood volumes for research, patients with weight <4kg will be excluded.
* Patients will not be excluded on the basis of gender, ethnicity, genetic diagnosis, gestational age at birth, non-cardiac comorbidity, or pre-operative medication regimen.

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with single ventricle heart disease undergoing trans-catheter evaluation in anticipation of superior cavo-pulmonary anastomosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in ET1 concentration between controls, study patients at pre-SCPA catheterization, and study patients in the post-operative period. | 48 hours post-operatively
Difference in metabolomics profile between controls, study patients at pre-SCPA catheterization, and study patients in the post-operative period. | 48 hours post-operatively

SECONDARY OUTCOMES:
Association between ET1 concentration at pre-SCPA catheterization in study patients and clinical metrics of pre-operative pulmonary adequacy. | 48 hours post-operatively
Association between metabolomics profile in study patients and clinical metrics of pre-operative pulmonary adequacy. | 48 hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Frank, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frank BS, Khailova L, Silveira L, Mitchell MB, Morgan GJ, Hsieh EWY, DiMaria MV, Twite M, Klawitter J, Davidson JA. Proteomic profiling identifies key differences between inter-stage infants with single ventricle heart disease and healthy controls. Transl Res. 2021 Mar;229:24-37. doi: 10.1016/j.trsl.2020.10.001. Epub 2020 Oct 9. PMID 33045409